CLINICAL TRIAL: NCT05903859
Title: Improvement of Reproductive Function in Men With Spinal Cord Injury (SCI)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emad Ibrahim, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20230188; SC220060 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Infertility, Male
Keywords: Spinal cord injury
MeSH Terms: conditions — Infertility, Male; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Full dose group (Experimental): Participants in this group will receive the full dose of probenecid for a total of 90 days.
  Interventions: Drug: Probenecid 500 Milligrams (mg)
- Half dose group (Experimental): Participants in this group will receive half the dose of probenecid for a total of 90 days.
  Interventions: Drug: probenecid 250 Milligrams (mg)
- Control-placebo group (Placebo Comparator): Participants in this group will receive a placebo dose (No active ingredient) for a total of 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probenecid 500 Milligrams (mg) — Participants in this group will receive 500 mg of probenecid by mouth twice a day for a total of 90 days.
  Arms: Full dose group
Drug: probenecid 250 Milligrams (mg) — Participants in this group will receive 250 mg of probenecid by mouth twice a day for a total of 90 days.
  Arms: Half dose group
Drug: Placebo — Participants in this group will receive a placebo pill by mouth twice a day for a total of 90 days.
  Arms: Control-placebo group

SUMMARY:
This is a study of infertility which often occurs in men with spinal cord injury. Most men with spinal cord injury have a normal sperm count but abnormally low sperm motility - which means that the sperm does not swim well. This study will determine if a medicine given by mouth will improve sperm motility in men with spinal cord injuries. The medicine is called probenecid.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a traumatic spinal cord injury.
2. Subject is male and is 18 years or older.

Exclusion Criteria:

1. Subject has been injured less than 1 year.
2. The subject is known to be azoospermic.
3. The subject has an indwelling urethral Foley catheter.
4. Subject is under the age of 18 years.
5. Subject has an unstable medical condition including, but not limited to, Crohn's disease, ulcerative colitis, colon cancer or has other conditions deemed to be exclusionary per the Investigator.
6. Subject is unable to consent or comprehend the procedures and their implications.
7. Subject has a permanent implanted electrical device, i.e., cardiac pacemaker, phrenic nerve stimulator, spinal cord stimulator, etc.
8. Any subject for whom the procedure or medication is otherwise contraindicated.
9. Subject has hypersensitivity to probenecid.
10. Subject has a history of uric acid kidney stones and/or peptic ulcer.
11. The subject has had a febrile Urinary Tract Infection (UTI) within the 2 months prior to enrollment.
12. The subject is taking methotrexate, aspirin, other salicylates, or anti-inflammatory medicines.
13. The subject has a history of Glucose-6-phosphate dehydrogenase (G6PD) deficiency.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in total motile sperm count | Baseline, up to 6 months post intervention, up to 6 months post follow up.
  The total sperm count will be assessed by calculating semen volume times sperm count times sperm motility percentage.The unit of measurement is in Millions.

SECONDARY OUTCOMES:
Change in percentage sperm DNA fragmentation | Baseline, up to 6 months post intervention, up to 6 months post follow up.
  The percentage of DNA fragmented sperm in specimen
Change in percentage of sperm viability | Baseline, up to 6 months post intervention, up to 6 months post follow up.
  The percentage of viable sperm ion specimen
Change in semen inflammasome markers | Baseline, up to 6 months post intervention, up to 6 months post follow up.
  Markers will be measured in picogram/milliliter units
Number of treatment-related adverse events | Up to 6 months post follow up.
  Treatment-related adverse events will be assessed by the treating physician using Common Terminology Criteria for Adverse Events 4 (CTCAE 4)

CONTACTS AND LOCATIONS:
Overall Officials: Emad Ibrahim, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ibrahim E, Aballa TC, Lynne CM, Brackett NL. Oral probenecid improves sperm motility in men with spinal cord injury. J Spinal Cord Med. 2018 Sep;41(5):567-570. doi: 10.1080/10790268.2017.1320875. Epub 2017 May 2. PMID 28464732